CLINICAL TRIAL: NCT03498534
Title: Evaluation of the Impact of Diabetes Control on Transmission and Development of Tuberculosis in the General Population
Brief Title: Evaluation of Diabetes Control and Effect on Transmission and Development of Tuberculosis
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Due to administrative procedures
Sponsor: Instituto Nacional de Salud Publica, Mexico (Other)
Responsible Party: Principal Investigator, Ma. de Lourdes Garcia Garcia, Director of the Center of Research in Infectious Diseases, Instituto Nacional de Salud Publica, Mexico
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CI-543
Record Dates: First submitted 2012-03-28; First posted 2018-04-13 (Actual); Last update posted 2018-04-17 (Actual); Status verified 2018-04

CONDITIONS: Latent Tuberculosis; Diabetes Mellitus
Keywords: Treatment; Latent infection; Tuberculosis; Interferon gamma
MeSH Terms: conditions — Latent Tuberculosis; Diabetes Mellitus; Latent Infection; Tuberculosis | interventions — Isoniazid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Patients with a -TST (Active Comparator): In all patients with a negative TST test, Isoniazid 300 mg per day will be administered for 6 months
  Interventions: Drug: Isoniazid 300Mg Tab
- Patients with a +TST (Active Comparator): In patients with a +TST test researchers will test for HIV, hepatic function and we will take a chest x-ray. Isoniazid 300 mg per day will be administered for 6 months
  Interventions: Drug: Isoniazid 300 MG
- HIV positive patients (Active Comparator): The researchers will test hepatic function and take a chest x-ray. Isoniazid 300 mg per day will be administered for 6 months
  Interventions: Drug: Isoniazid 300 MG

INTERVENTIONS:
Drug: Isoniazid 300Mg Tab — -TST tests will receive isoniazid 300Mg Tab for 6 months
  Other Names: Isoniazid 300 mgs.
  Arms: Patients with a -TST
Drug: Isoniazid 300 MG — + TST test will receive isoniazid 300MG Tab for 6 months
  Other Names: Isoniazid
  Arms: Patients with a +TST
Drug: Isoniazid 300 MG — HIV positive patient will receive isoniazid 300MGTab for 6 months
  Other Names: Isoniazid 300 mg per day
  Arms: HIV positive patients

SUMMARY:
Clinical test (essay) randomized to evaluate the toxicity adherence and efficiency of the chemoprophylaxis of tuberculosis (TB) in subjects with Diabetes Mellitus (DM) and latent TB. (600 subjects followed(continued) by 15 months). 3rd stage. Patients with DM and TB will be included to determine if the strict control of the dm achieved in clinics of the first level of attention improves clinical manifestations of tb, the result of treatment, the frequency of relapses, the mortality and the transmission to contacts.

Elispot will be used to measure TB development and the time for the bacteriological negativization and biochemical parameters as well as tuberculin skin test (TST), quantiferon, in contacts. (160 patients 600 contacts followed(continued) for 12 months). additional there will be evaluated the socioeconomic impact of both diseases and his(her) control. 1er year: transverse study and recruitment years 2 and 3 participants' follow-ups in clinical tests(essays).

ELIGIBILITY:
Inclusion Criteria:

* Positive HIV TST tuberculin

Exclusion Criteria:

* Previous TB treatment Hepatic failure AIDS

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-09; Primary Completion 2012-12 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Development of active TB | 6 months
  Researchers will test patients at day 0 and day 180 of treatment to detect the development of active TB

CONTACTS AND LOCATIONS:
Overall Officials: Garcia-Garcia Lourdes, Doctor, Principal Investigator — National Institute of public Health